CLINICAL TRIAL: NCT02661867
Title: Pelvic Floor Function Evaluation of Singleton Primiparae After Vaginal Delivery and Cesarean Section: Seven to Twelve-Year Long Observational Cohort Study
Brief Title: Pelvic Floor Function Evaluation of Singleton Primiparae After Vaginal Delivery and Cesarean Section
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Martin Huser, doctor, Brno University Hospital
Other Study IDs: Plure
Record Dates: First submitted 2016-01-16; First posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Pelvic Floor Disorders
Keywords: Childbirth; Pelvic organ prolapse; Urinary incontinence; Fecal incontinence
MeSH Terms: conditions — Pelvic Floor Disorders; Pelvic Organ Prolapse; Urinary Incontinence; Fecal Incontinence | interventions — Parturition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VD: Vaginal delivery group - women who gave birth of offspring through the vagina without the use of special instruments such as forceps or a vacuum extractor (instrumental vaginal delivery)
  Interventions: Behavioral: delivery
- CS: Cesarean section group - women delivered by surgical procedure in which one or more incisions are made through a mother's abdomen and uterus to deliver a baby. Cesarean section is performed when a vaginal delivery would put the baby's or mother's life or health at risk.
  Interventions: Behavioral: delivery

INTERVENTIONS:
Behavioral: delivery — delivery either vaginal or by cesarean section

SUMMARY:
Objective of this longitudinal observational cohort study was to analyze incidence of pelvic floor dysfunction (PFD) symptoms, including pelvic organ prolapse (POP), urinary incontinence (UI), and fecal incontinence (FI), seven to twelve years after delivery, in two groups of singleton primiparae after vaginal delivery (VD) and cesarean section (CS).

DETAILED DESCRIPTION:
Pelvic floor disorders (PFD) usually refers to three definable groups of symptoms that include pelvic organ prolapse (POP), urinary incontinence (UI), and fecal incontinence (FI). The prevalence of these conditions increases with age, but in general, PFD affect 20-50 % of women throughout their lives. Thus, PFD are common and have significant societal impact. Another important PFD risk factor is childbearing. Specifically, these disorders are more common among multiparas. Vaginal delivery (VD) has been considered the main contributing factor because of pelvic floor muscle, fascia, and nerves damage.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* cephalic presentation
* delivery in term (gestational week 38-42)
* no other childbirth during study period

Exclusion Criteria:

- operative vaginal delivery (vacuum extraction or forceps delivery)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primiparae delivered vaginally (VD group) or by cesarean section (CS group) during the years 2002-2007 in university-based large perinatology center
Sampling Method: Probability Sample
Enrollment: 865 (Actual)
Dates: Start 2002-01; Primary Completion 2007-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pelvic organ prolapse symptoms score | seven years after delivery
  calculated from validated questionnaire International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF)

SECONDARY OUTCOMES:
Urinary incontinence symptoms score | seven years after delivery
  calculated from validated questionnaire Pelvic Organ Prolapse Distress Inventory (POPDI-6)
Fecal incontinence symptoms score | seven years after delivery
  calculated from validated questionnaire Wexner Fecal Incontinence Score (WS)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Memon H, Handa VL. Pelvic floor disorders following vaginal or cesarean delivery. Curr Opin Obstet Gynecol. 2012 Oct;24(5):349-54. doi: 10.1097/GCO.0b013e328357628b. PMID 22907482
- [Derived] Huser M, Janku P, Hudecek R, Zbozinkova Z, Bursa M, Unzeitig V, Ventruba P. Pelvic floor dysfunction after vaginal and cesarean delivery among singleton primiparas. Int J Gynaecol Obstet. 2017 May;137(2):170-173. doi: 10.1002/ijgo.12116. Epub 2017 Mar 1. PMID 28171703